CLINICAL TRIAL: NCT00110708
Title: A Randomized, Placebo-Controlled Phase II Trial Evaluating Safety and Efficacy of Oral Human Immunoglobulin in the Treatment of Gastrointestinal Dysfunction Associated With Autistic Disorder in Pediatric Patients From 2 to 18 Years of Age
Brief Title: Safety and Efficacy Study in the Treatment of Intestinal Problems Associated With Autism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PediaMed Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol 004
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Autism; Autistic Disorder; Child Development Disorders, Pervasive; Gastrointestinal Diseases; Signs and Symptoms, Digestive
Keywords: autism; gastrointestinal dysfunction; autistic disorder; diarrhea; constipation; abdominal pain; gastrointestinal problems associated with autism; immune globulin; immunoglobulin; Immunoglobulins, Intravenous; Intestinal Mucosa/immunology/pathology; Administration, Oral; Autistic Disorder/*drug therapy; Child Behavior/*drug effects; Constipation/drug therapy; Diarrhea/drug therapy; Gastrointestinal Agents/*therapeutic use
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive; Gastrointestinal Diseases; Signs and Symptoms, Digestive; Diarrhea; Constipation; Abdominal Pain | interventions — Immunoglobulins, Intravenous

INTERVENTIONS:
Drug: Oralgam (human immunoglobulin)

SUMMARY:
The purpose of this study is to determine if human immunoglobulin given by mouth twice a day is effective in treating the persistent gastrointestinal (GI) problems such as diarrhea, constipation, abdominal pain, and bloating, in children with autism.

DETAILED DESCRIPTION:
Autistic GI Dysfunction (AGID) is a term that describes a constellation of GI signs and symptoms often found in children with autistic disorder, including abdominal pain, constipation, chronic diarrhea, alternating constipation and diarrhea, gaseousness, bloating, and reflux.

The objective of this study is to assess the potential efficacy of oral immunoglobulin in reducing a wide range of GI symptoms in children and adolescents diagnosed with autistic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 2 years to 18 years of age (up to, but not inclusive of the 18th birthday)
* Diagnosis of autistic disorder corroborated by an Autism Diagnostic Interview - Revised (ADI-R) assessment performed by a certified investigator
* Physician Clinical Global Impression of Severity (of Autistic Disorder)
* History of chronic, persistent gastrointestinal disturbance
* No elective changes in medication, diet intervention, or behavioral therapy during the study (18 weeks total)

Exclusion Criteria:

* Evidence of a gastrointestinal infection or GI abnormality
* A known diagnosis of other gastrointestinal pathology
* Antibiotic and/or antifungal (e.g. nystatin) medication
* Chelation therapy
* Medication affecting gastrointestinal transit
* Planned use of prohibited drugs or agents that could affect GI transit
* Changes in diet intervention within 30 days prior to the screening visit
* Changes in alternative medical therapies or dietary supplements within 30 days prior to the screening visit
* Adding and/or changing behavior modification or psychotherapy during participation in the study
* Adding or changing psychotropic medication during participation in the study
* DSM-IV diagnosis of a pervasive developmental disorder other than autistic disorder
* Evidence of a seizure disorder, diagnosis of fragile X syndrome, tuberous sclerosis complex, liver disease, pancreatic disease, cystic fibrosis, or chronic infection
* Previous gastrointestinal surgery
* Pregnancy
* Participation in another investigational study
* Significant deviation from normal laboratory test values at baseline
* IgA deficiency (serum IgA < 5 mg/dL)
* A history of severe hypersensitivity to human immunoglobulin
* Treatment with any human immunoglobulin and/or immunoglobulin products
* Any concurrent medication that would compromise subject's tolerance of drug or compliance with the protocol

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2005-04; Study Completion 2006-06

PRIMARY OUTCOMES:
Global improvement in gastrointestinal function

SECONDARY OUTCOMES:
Assessment of behavior (improvement and severity); additional assessments of gastrointestinal conditions

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Center for Autism Research and Education, Phoenix, Arizona
  - University of California Davis, MIND Institute, Sacramento, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - University of Florida HSC, Gainesville, Florida
  - International Child Development Resource Center, Melbourne, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Developmental Disabilities Center, Kansas City, Kansas
  - Bluegrass Clinical Research, Louisville, Kentucky
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Hardy Health Associates, Hingham, Massachusetts
  - Pivotal Research Centers - Detroit, Royal Oak, Michigan
  - Mercy Health Research, St Louis, Missouri
  - Robert Wood Johnson Medical School, Piscataway, New Jersey
  - Strong Center for Developmental Disabilities, University of Rochester Medical Center, Rochester, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nisonger Center Ohio State University, Columbus, Ohio
  - Merck Child Outpatient Clinic, Pittsburgh, Pennsylvania
  - North San Antonio Healthcare Associates, San Antonio, Texas
  - Autism Spectrum Treatment and Research Center, Seattle, Washington

REFERENCES:
- [Derived] Handen BL, Melmed RD, Hansen RL, Aman MG, Burnham DL, Bruss JB, McDougle CJ. A double-blind, placebo-controlled trial of oral human immunoglobulin for gastrointestinal dysfunction in children with autistic disorder. J Autism Dev Disord. 2009 May;39(5):796-805. doi: 10.1007/s10803-008-0687-y. Epub 2009 Jan 16. PMID 19148734